CLINICAL TRIAL: NCT01341730
Title: Evaluation of the Effect of Atorvastatin and Pioglitazone in Carotid Atherosclerosis With the Use of 18Fluoride-Fludeoxyglucose(FDG) Positron Emission Tomography-computed Tomography (PET-CT)Imaging
Brief Title: The Effect of Atorvastatin and Pioglitazone on Carotid Atherosclerosis With the Use of Positron Emission Tomography-computed Tomography (PET-CT)
Acronym: PIONEER
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Collaborators: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Eun Ho Choo, Cardiovascular Center, Seoul St. Mary's Hospital,, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CUKCVC
Record Dates: First submitted 2011-04-20; First posted 2011-04-26 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Atherosclerosis; Coronary Artery Disease
Keywords: Atherosclerosis; Pioglitazone; Atorvastatin; PET CT
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease | interventions — Atorvastatin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin 20 mg (Active Comparator): After the subject take PET CT, he or she is randomized to either " Atorvastatin 20 mg" group or " Atorvastatin 20 mg+ Pioglitazone 30 mg". The " Atorvastatin 20 mg" group is to take atorvastatin 20 mg and take follow up PET CT in 3 months
  Interventions: Drug: Atorvastatin 20mg
- Atorvastatin 20 mg + Pioglitazone 30 mg (Experimental): After the subject take PET CT, he or she is randomized to either " Atorvastatin 20 mg" group or " Atorvastatin 20 mg+ Pioglitazone 30 mg". The " Atorvastatin 20 mg + Pioglitazone 30 mg" group is to take atorvastatin 20 mg + pioglitazone 30 mg and take follow up PET CT in 3 months
  Interventions: Drug: Atorvastatin 20 mg + Pioglitazone 30 mg

INTERVENTIONS:
Drug: Atorvastatin 20mg — 20 mg QD for 3 months
  Other Names: Lipitor 20mg
  Arms: Atorvastatin 20 mg
Drug: Atorvastatin 20 mg + Pioglitazone 30 mg — atorvastatin 20 mg plus pioglitazone 30 mg QD for 3 months
  Other Names: Lipitor 20mg plus Actos 30mg
  Arms: Atorvastatin 20 mg + Pioglitazone 30 mg

SUMMARY:
This study is a prospective randomized clinical trial and to compare the antiinflammatory effect of atorvastatin single therapy and atorvastatin and pioglitazone combination therapy in carotid arteries of stable and unstable angina patients by PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* The subject who has undergone percutaneous coronary intervention due to coronary artery disease ( stable angina or unstable angina)
* The subject described above who has atherosclerotic plaque in his/her carotid artery by carotid ultrasonography
* The subject who or a legal representative agrees to the clinical trial and gives written permission to the IRB-approved form.

Exclusion Criteria:

* The subjets who have taken statins or thiazolidinedione with 4 weeks
* Marked elevated liver enzyme ( more than 2.5 fold compared to reference range)
* Renal insufficiency patients ( serum creatinine more than 2 mg/dl)
* Congestive heart failure ( NYHA class 2-4)
* Acue myocardial infarction
* Unstable angina with ST segment deviation
* Pregnancy
* The subjects enrolled in another studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kiyuk Chang, M.D., Principal Investigator — Department of Medicine, Seoul St. Mary's hospital, The Catholic University of Korea, Colege of Medicine
Locations (1):
- Cardiovascular center, Seoul St. Mary's hospital, Seoul, South Korea

REFERENCES:
- [Derived] Choo EH, Han EJ, Kim CJ, Kim SH, O JH, Chang K, Seung KB. Effect of Pioglitazone in Combination with Moderate Dose Statin on Atherosclerotic Inflammation: Randomized Controlled Clinical Trial Using Serial FDG-PET/CT. Korean Circ J. 2018 Jul;48(7):591-601. doi: 10.4070/kcj.2017.0029. PMID 29968431

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated prematurely due to slow enrollment.
Period: Overall Study
Arm/Group | Atorvastatin 20 mg | Atorvastatin 20 mg + Pioglitazone 30 mg
Started | 20 | 21
Completed | 16 | 17
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Population: Four patients from each group withdrew the consent after enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin 20 mg | Atorvastatin 20 mg + Pioglitazone 30 mg | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (11.0) | 63.4 (10.5) | 63 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 8 | 12 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 17 | 33
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Difference of Standardized Uptake Value (SUV) of Atherosclerotic Plaque in Carotid Artery by PET CT
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: standardized uptake value (SUV)
Arm/Group | Atorvastatin 20 mg | Atorvastatin 20 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 16 | 17
standardized uptake value (SUV) | -0.06 (0.04) | -0.10 (0.07)

2. Secondary Outcome: Difference PET CT Parameters in 3 Months Compared to Initial Evaluation
Description: Change of Maximum Standardized Uptake Value (SUVmax),Mean Standardized Uptake Value (SUVmean)- no unit for this value
Time Frame: 3 months
Population: Data were not collected
Groups:
- Atorvastatin 20 mg; Atorvastatin 20 mg + Pioglitazone 30 mg: Data were not collected
Arm/Group | Atorvastatin 20 mg | Atorvastatin 20 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Difference of Laboratory Data Compared to Initial Evaluation
Description: Change of high sensitivity C-reactive protein (hsCRP, mg/dl) Change of low density lipoprotein cholesterol(mg/dl) Change of high density lipoprotein cholesterol(mg/dl) Change of triglyceride (mg/dl) Change of matrix metalloproteinase 9 (mcg/ml) Change of plasminogen activator inhibitor (PAI)-1 (ng/ml) Change of Homeostatic Model Assessment (HOMA) index (%)
Time Frame: 3 months
Reporting Status: Not Posted

4. Secondary Outcome: Clinical Incidents
Description: Major adverse cerebro-cardiovascular event: a composite of cardiac death, nonfatal myocardial infarction, stroke, and target vessel revascularization
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Atorvastatin 20 mg | Atorvastatin 20 mg + Pioglitazone 30 mg
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No